CLINICAL TRIAL: NCT06007885
Title: Examining Capacity Building of Youth With Physical Disabilities to Pursue Participation Following the Pathways and Resources for Engagement and Participation (PREP) Intervention. An Individual-based Mixed Methods Study.
Brief Title: Examining Capacity Building of Youth With Physical Disabilities to Pursue Participation Following the PREP Intervention.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dana Anaby, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-50-2023-1824
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Spinal Cord Injuries; Spina Bifida; Musculoskeletal Disorder; Juvenile Arthritis; Amputation; Cerebral Palsy
Keywords: participation; environmental barriers; youth; disabilities; capacity building
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Dysraphism; Musculoskeletal Diseases; Arthritis, Juvenile; Cerebral Palsy | interventions — Health Resources

STUDY DESIGN:
Intervention Model Description: A 26-week individual-based convergent mixed methods design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-based activity program (Experimental): Engagement in 8-week community-based activity program.
  Interventions: Other: Pathways and Resources to Engagement and Participation (PREP)

INTERVENTIONS:
Other: Pathways and Resources to Engagement and Participation (PREP) — Participants engage in an 8-week community-based activity of their choice (Goal#1). To engage in the selected activity, an Occupational Therapist (OT) will meet with each youth in their home/community and use the PREP 5 steps (Make goals; Map out a plan; Make it happen; Measure the process and outcomes; Move forward). The OT will work with the youth to search for the programs, identify and remove potential environmental barriers for participation (e.g., accessibility, equipment) and educate instructors regarding the youth's specific needs. This process, which includes up to 9 hours of OT support, will set the stage for enrolment of the youth in a community activity for a period of 8 weeks. The intervention will be repeated for a new goal (Goal#2). However, for Goal#2, youth will have the opportunity to select and pursue their new goal (#2) for 8 weeks without OT support first. Then, the OT will provide the PREP intervention for up to 6 weeks to achieve Goal #2.
  Other Names: Pathways and Resources for Engagement and Participation (PREP)

SUMMARY:
The goal of this clinical trial is to learn about how a participation-based intervention builds capacity of youth with physical disabilities to pursue activities of their choice in the community. The investigators plan to examine in what ways working with a therapist to set up and engage in an 8-week self-chosen community-based activity builds capacity of youth with physical disabilities to pursue a new activity of their choice in the community without the support of a therapist.

During this study, participants will be followed for 26 weeks. Youth will work with an occupational therapist (OT).

* In the first week, the OT will meet with youth to set a community-based leisure goal. Examples of activities could include music, sports, cooking lessons, painting, or photography, in the youth's community.
* The OT will work with youth to identify and remove barriers. They will also adapt the activity to help youth do the activity for 8 weeks. During this time, the OT will perform site visits to consult and support youths' involvement as needed. (Weeks #1-8)
* Youth will have a four-week break after completing their first activity. (Weeks #9-12). Then, youth will be asked to choose a second (new) activity. They will try to start this activity for 8 weeks without the OT. (Weeks #13-20)
* At the end of these 8 weeks, the same therapist will help the youth for 6 weeks if needed to do their second activity. (Weeks #21-26)

Youth will be asked to complete the following online:

1. A standard demographic questionnaire (during the first meeting).
2. Rate their perceived performance in the chosen activity once a week.
3. A questionnaire about their daily participation in the community. This will be done at the start and end of the study.
4. A questionnaire about how well they feel they are able to do things. This will be done three times.
5. Share steps they take to participate in the activity. This will be done through a weekly diary entry. In addition, three one-on-one interviews (for about an hour each) will be done remotely (using Microsoft TEAMS) to share their experience pursuing their selected activities. Interviews will be done before starting their second (new) activity, after 8 weeks of pursuing the new activity on their own, and after 6 weeks with OT support. These interviews will be video, and audio recorded and transcribed.

This study examines 'real-life' experiences and participation outcomes of youth with physical disabilities after a participation-based capacity-building intervention.

DETAILED DESCRIPTION:
Participation of youth with disabilities is severely restricted by environmental barriers, leading to poorer transition outcomes as compared to their peers without disabilities. In pediatric rehabilitation, capacity building - a process encompassing change in knowledge and skills focusing on future growth and development of the client's potential - is necessary for creating sustainable change toward participation outcomes. Building capacity of youth to develop and use solution-based strategies in new contexts is critical for making a successful transition to adulthood. The PREP (Pathways and Resources to Engagement and Participation) is one example of a participation-based intervention that aims to build capacity of youth to solve problems through removing environmental barriers and building support for participation in a 'real-world' context. PREP, which includes 5 standardized steps, i.e., Make goals; Map out a plan; Make it happen; Measure the process and outcomes; and Move forward, has been shown to significantly improve participation in self-chosen activities of youth with physical disabilities ages 12-25. However, outcomes related to building capacity of youth to problem-solve and pursue sustainable participation beyond the support of a therapist have not been evaluated. This study addresses the gap in knowledge by exploring 'real-life' experiences and participation outcomes of youth with physical disabilities after a participation-based capacity-building intervention.

This study aims to understand in what ways the PREP intervention builds capacity of youth with physical disabilities to pursue participation in new self-chosen activities. The main questions it aims to answer are: 1) What are the experiences of youth with physical disabilities as they pursue a new self-chosen activity (goal #2) for 14 weeks (8-weeks independently, and 6-weeks with OT support), starting 4 weeks after completion of the initial PREP intervention (goal #1)?; 2) To what extent does youth's participation in a new self-chosen activity (goal #2) change over 14 weeks of pursuing the new activity (8-weeks independently, and 6-weeks with OT support) in terms of trend and level, starting 4 weeks following completion of the initial PREP intervention for goal#1? and 3) How do youth's experiences pursuing participation in a self-chosen activity following the intervention relate to data measuring levels of participation in the new activity over time, while also considering youth's levels of self-determination and overall community participation profiles?

A 26-week individual-based convergent mixed methods design will explore the capacity building process and outcomes following the completion of the PREP intervention. Ten youth with physical disabilities (ages 15-24), will complete the PREP for one goal with the therapist for 8 weeks. Four weeks after completion, youth will work independently toward a new goal for 8 weeks, after which they will be supported by a therapist for an additional 6 weeks if needed to achieve their new goal.

Youth will be interviewed at three time points to explore their experiences working towards their new goal (QUAL). Youth will document the process (i.e., strategies, challenges) of pursuing their new goal through a weekly PREP diary over 14 weeks (QUAL). Changes in participation levels for goals are measured weekly using the COPM over 8 weeks (goal#1) and 14 weeks (8 weeks without the therapist and 6 weeks with therapist support for goal#2) (QUAN). The resulting 20 trajectories of change (10 for goal#1 and 10 for goal #2) are analyzed visually for trend and level. To complement COPM data collected for the new goal, the weekly PREP diary, completed over the 14 weeks, will undergo inductive content analysis and will be used to describe youth's participation over time providing context about the trends and levels observed for each youth's pursuit of their new activity (QUAL). The 30 transcripts (10 youth x 3 interviews) are analyzed using inductive reflexive thematic analysis. Data collected from all sources (COPM, diary, interviews) is triangulated to account for the process of capacity building and its outcomes. A joint display organized by participant will be used for a side-by-side comparison of quantitative and qualitative results. An iterative process will be used to compare results within and across participants to look for potential inconsistencies or complementary findings between the sets of data. Meta-inferences are generated by comparing QUAN (COPM score/trajectories) and QUAL data (interviews and diary entries). The meta-inferences generated through the joint display and additional insights will be discussed using a narrative approach. Data will also be collected to describe the sample of youth in terms of their current community participation profiles (using the Youth, Young-adult Participation and Environment Measure; Y-PEM) and self-reported levels of self-determination (using the American Institutes for Research - Student Self-Determination Scale; AIR-S). Detailed information about the participants can inform how the intervention is applicable to different individuals, thus supporting the uptake of research into practice.

The research team includes 4 international and interdisciplinary experts from the fields of occupational therapy, social work, and psychology, all with extensive knowledge in participation-based interventions as well as experience conducting complex clinical trials. This project also involves intersectoral partnerships with managers/local decision-makers from both the clinical and non-clinical communities who all have a special interest (and knowledge) in transitioning of youth with physical disabilities to adult roles and adult care. With diverse backgrounds including rehabilitation services, social and recreation organizations (from both public and non-profit sectors), and individuals with lived experience of disability, these partners form a rich consultative committee to advise the project.

This study will contribute evidence towards the long-term impacts following a participation-based capacity building intervention for youth with physical disabilities. Additionally, this study will contribute to our understanding of the elusive yet important construct of capacity-building. Such new knowledge may advance methods for evaluating efficiency of participation-focused interventions and may be of interest to both clinicians and decision-makers.

ELIGIBILITY:
Inclusion Criteria:

* have a physical disability (e.g., cerebral palsy, spina bifida, musculoskeletal disorders)
* restricted mobility, such as an inability to navigate all surfaces and stairs independently and safely without the use of aids, physical assistance or external support

Exclusion Criteria:

* have previously received the PREP intervention
* severe intellectual disabilities and/or complex communication issues (due to the demands of completing questionnaires/diaries and interviews).

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Weekly for 8 weeks Goal #1; Weekly for 14 weeks Goal #2
  A gold-standard 10-point scale that measures activity performance. Score ranges from 1 (unable to perform) to 10 (performs extremely well)

SECONDARY OUTCOMES:
AIR Self-Determination Scale (Student Form) | 3x (Week 1-baseline, Week 12-before starting goal#2, Week 26-end of study)
  The AIR-S profile is divided into four sections (6 items in each, rated on a 5-point scale) which make up two subscale scores: ability ('Things I do') and perception ('How I Feel') together provide a capacity score at home ('What Happens at Home') and school ('What Happens at School') provide an opportunity score. An overall percentage (out of 100%) for level of self-determination is determined if all sections are completed and can be used to compare within the individual across time. Scores within the capacity and opportunity subcategories can also be compared descriptively since the self-determination process is broken down into thinking-doing-adjusting.
Youth, Young-adult Participation and Environment Measure (Y-PEM) - Community Domain | 2x (Week 1-baseline, Week 26-end of study)
  Self-reported participation-based measure capturing important aspects of participation.
  Y-PEM Scales: Frequency (never = 0 to daily = 7); Involvement (minimally involved = 1 to very involved = 5); Desire for Change 1. No or yes, if yes, youth identify a) where change is desired (frequency, involvement, and/or variety), and b) be more/less involved; Features of the Environment (1= Usually makes harder, 2= Sometimes helps, sometimes makes harder, 3= Usually helps, 4= Not an issue); Perceived Adequacy / Availability of Resources (1= usually no, 2= sometimes yes, sometimes no, 3= usually yes, 4= not needed)

OTHER OUTCOMES:
Individual Semi-Structured Interviews | 3x (Week 12-before starting goal#2, Week 20-after 8 weeks independently pursuing goal#2, Week 26-after 6 weeks with therapist support for goal#2/end of study)
  Three 1-hour semi-structured interviews will be completed with each youth to explore their experiences pursuing participation in a new activity after the initial PREP intervention. Specifically, an interview guide comprised of 12 open-ended questions will be used.
Electronic PREP Diary | Weekly for 14 weeks (goal #2)
  Structured activity log reflecting elements of the PREP Forms (e.g., environmental barriers, supports, and strategies) where youth will document actions they take towards pursuing a new goal over 14 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Anaby, PhD, Principal Investigator — McGill University
Locations (1):
- Lethbridge-Layton-Mackay Rehabilitation Center of CIUSSS West-Central Montreal (Mackay site), Montreal, Quebec, Canada